CLINICAL TRIAL: NCT06019169
Title: Randomized Pilot Trial: Impact of YOGA on the Quality of Life and Well-being of Heart Failure Patients
Brief Title: Impact of YOGA on the Quality of Life and Well-being of Heart Failure Patients
Acronym: YOG-IC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP230227
Record Dates: First submitted 2023-08-17; First posted 2023-08-31 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-08

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart Failure; Yoga; randomized; SF36

STUDY DESIGN:
Intervention Model Description: Pilot study, prospective, monocentric controlled in open label, Randomization ratio 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workshops around social activities (Active Comparator): Participate in workshops around social activities. 4 sessions are planned (2 face-to-face and 2 remotely) per month for 3 months.
  Interventions: Other: storytelling activities
- Yoga classes (Experimental): Participation in YOGA classes performed by Mme Laura BOGANI from The Blue Fish LAB Association. There are 4 sessions of 45 minutes (2 face-to-face and 2 remote) per month for 3 months.
  Interventions: Other: Yoga arm

INTERVENTIONS:
Other: Yoga arm — Participation in YOGA classes performed by Mme Laura BOGANI from The Blue Fish LAB Association. There are 4 sessions of 45 minutes (2 face-to-face and 2 remote) per month for 3 months. An attendance sheet will be completed at each session.
  Arms: Yoga classes
Other: storytelling activities — Participate in workshops around storytelling led by the association of storytellers l'Age D'or. 4 sessions are planned (2 face-to-face and 2 remotely) per month for 3 months. An attendance sheet will be completed at each session.
  Arms: Workshops around social activities

SUMMARY:
Heart failure (HF) is a chronic disease that has a strong impact on quality of life and is often accompanied by anxiety and depression symptoms that can contribute to poor treatment compliance. The overall management of heart failure is currently part of the recommendations and, alongside drug therapy and electrical devices that can be proposed, lifestyle changes (diet, physical activity) can help improve well-being. and perhaps patient prognosis. Yoga is an ancient practice, known to improve the emotional and physical well-being of individuals. There is no formal medical contraindication to this practice, which can be perfectly adapted to the patient's condition. However, very few patients with heart failure practice yoga. A few randomized trials with small numbers as well as the combined analysis of several studies have shown the benefit of yoga in heart failure. The main objective of the research is to demonstrate the improvement in the quality of life induced by the regular practice of yoga in the management of stabilized chronic heart failure patients. Secondly, we will evaluate the effectiveness of regular yoga practice on improving the clinical condition of chronic heart failure patients.

DETAILED DESCRIPTION:
Study design :

Pilot study, prospective, monocentric controlled in open, Randomization ratio 1:1: in two parallel groups

* Arm control workshops around social activities
* Yoga arm (Y): Participation in YOGA classes. There are 4 sessions of 45 minutes (2 face-to-face and 2 remote) per month for 3 months. An attendance sheet will be completed at each session.

Population concerned :

Patients with stabilized chronic heart failure (last episode of acute heart failure dating back more than a month) followed at the Pitié Salpêtrière cardiology institut

The study may be offered to any stabilized heart failure patient followed in the study centre. Visit V1 (D0): Information, Inclusion and randomization Visit V2 (M3): final visit. Between V1 and V2: weekly workshop sessions around storytelling (arm C) or Hatha yoga (Arm Y).

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years old
* Chronic heart failure patient defined by: Most recent LVEF ≤50% (regardless of measurement method)
* Stabilized (last episode of acute heart failure dating back more than a month) in NYHA stage I to III dyspnoea, ambulatory, discharged from hospital for > 1 month
* Drug treatment optimized according to the judgment of the investigator
* Ability to participate in activities as proposed (remote or face-to-face)
* Patient affiliated with a social security scheme
* Written consent to participate

Exclusion Criteria:

* Patients who have practiced yoga regularly (> once a month) in the six months prior to selection.
* Current pregnancy / lactation
* Etiology of heart failure: hypertrophic cardiomyopathy, restrictive heart disease or severe curable valve disease
* Severe renal impairment GFR<25ml/min/1.73 m2 or on dialysis.
* Persons subject to legal protection measures (guardianship, curatorship)
* Person not "receptive" to the practice of yoga
* Participation in intervention research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2027-03-26 (Estimated); Study Completion 2027-04-26 (Estimated)

PRIMARY OUTCOMES:
SF-36 quality of life | at day 0 and maximum at 5 month
  The SF-36 quality of life self-questionnaire is one of the most widely used questionnaires to assess the quality of life of patients. Its result is between 0 and 100. It includes a physical summary score and a psychological summary score.

SECONDARY OUTCOMES:
Score Hospital Anxiety and Depression Scale (HAD) | at day 0 and maximum at 5 month
  Self questionnaire about nervous breakdown, min=0, max=42, higher score means a worse outcome
Weight (kg) | at day 0 and maximum at 5 month
  Weight measurement during the inclusion visit (1st visit) and at the last visit (2nd visit). we measure the delta between the 2 visits.
Waist circumference (cm) | at day 0 and maximum at 5 month
  Measurement of the waist circumference during the inclusion visit (1st visit) and at the last visit (2nd visit). we measure the delta between the 2 visits.
Heart rate (Bpm) | at day 0 and maximum at 5 month
  Measurement of the heart rate during the inclusion visit (1st visit) and at the last visit (2nd visit). we measure the delta between the 2 visits.
Blood pressure (mmHg) | at day 0 and maximum at 5 month
  Measurement of blood pressure during the inclusion visit (1st visit) and at the last visit (2nd visit). we measure the delta between the 2 visits.
NYHA assessment | at day 0 and maximum at 5 month
  Definition of the stage of heart failure by the NHYA classification at the inclusion visit (1st visit) and at the last visit (2nd visit). we measure the delta between the 2 visits.
Concentration of Nt-pro BNP Biomarker | 3 months before inclusion and maximum 7 months after inclusion
  Analysis of Nt-pro BNP biomarkers at the inclusion visit (1st visit) and at the last visit (2nd visit). we measure the delta between the 2 visits. They will be used to analyze the results of the assessments carried out according to the current practice of the center
Concentration of CRP Biomarkers | 3 months before inclusion and maximum 7 months after inclusion
  Analysis of CRP biomarkers at the inclusion visit (1st visit) and at the last visit (2nd visit). we measure the delta between the 2 visits. They will be used to analyze the results of the assessments carried out according to the current practice of the center
Concentration IL6 Biomarkers | 3 months before inclusion and maximum 7 months after inclusion
  Analysis of IL6 biomarkers during the inclusion visit (1st visit) and the last visit (2nd visit). we measure the delta between the 2 visits. They will be used to analyze the results of the assessments carried out according to the current practice of the center
Distance during 6-minute walk test | 3 months before inclusion and maximum 7 months after inclusion
  distance traveled by the patient in 6 minutes
Peak VO2 | 3 months before inclusion and maximum 7 months after inclusion
  Peak VO2 measurement on two different dates to analyze the results of walk tests carried out according to the center's current practice
VO2 charge level | 3 months before inclusion and maximum 7 months after inclusion
  VO2 charge level on two different dates to analyze the results of walk tests carried out according to the center's current practice
VE/VCO2 | 3 months before inclusion and maximum 7 months after inclusion
  Measurement of the VE/VCO2 ratio on two different dates to analyze the results of the walk tests carried out according to the current practice of the center
First ventilatory threshold | 3 months before inclusion and maximum 7 months after inclusion
  Measurement of the first ventilatory threshold on two different dates to analyze the results of the walking tests carried out according to the current practice of the center
First ventilatory load level | 3 months before inclusion and maximum 7 months after inclusion
  Measurement of the first ventilatory level of load on two different dates to analyze the results of the walking tests carried out according to the current practice of the center

CONTACTS AND LOCATIONS:
Overall Officials: Lise LEGRAND, Dr, Study Chair — Institut de Cardiologie - Hôpital La Pitié Salpêtrière (APHP); Gilles MONTALESCOT, Pr, Study Director — Institut de Cardiologie - Hôpital La Pitié Salpêtrière (APHP)
Locations (1):
- Institut de Cardiologie, Centre Hospitalier Universitaire Pitié Salpêtrière (APHP), UPMC, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aggarwal M, Bozkurt B, Panjrath G, Aggarwal B, Ostfeld RJ, Barnard ND, Gaggin H, Freeman AM, Allen K, Madan S, Massera D, Litwin SE; American College of Cardiology's Nutrition and Lifestyle Committee of the Prevention of Cardiovascular Disease Council. Lifestyle Modifications for Preventing and Treating Heart Failure. J Am Coll Cardiol. 2018 Nov 6;72(19):2391-2405. doi: 10.1016/j.jacc.2018.08.2160. PMID 30384895
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Pullen PR, Nagamia SH, Mehta PK, Thompson WR, Benardot D, Hammoud R, Parrott JM, Sola S, Khan BV. Effects of yoga on inflammation and exercise capacity in patients with chronic heart failure. J Card Fail. 2008 Jun;14(5):407-13. doi: 10.1016/j.cardfail.2007.12.007. Epub 2008 May 27. PMID 18514933
- [Background] Pullen PR, Seffens WS, Thompson WR. Yoga for Heart Failure: A Review and Future Research. Int J Yoga. 2018 May-Aug;11(2):91-98. doi: 10.4103/ijoy.IJOY_24_17. PMID 29755216
- [Background] Pullen PR, Thompson WR, Benardot D, Brandon LJ, Mehta PK, Rifai L, Vadnais DS, Parrott JM, Khan BV. Benefits of yoga for African American heart failure patients. Med Sci Sports Exerc. 2010 Apr;42(4):651-7. doi: 10.1249/MSS.0b013e3181bf24c4. PMID 19952833
- [Background] Diez-Quevedo C, Lupon J, Gonzalez B, Urrutia A, Cano L, Cabanes R, Altimir S, Coll R, Pascual T, de Antonio M, Bayes-Genis A. Depression, antidepressants, and long-term mortality in heart failure. Int J Cardiol. 2013 Aug 20;167(4):1217-25. doi: 10.1016/j.ijcard.2012.03.143. Epub 2012 Apr 14. PMID 22507552
- [Background] Snaith RP, Zigmond AS. The hospital anxiety and depression scale. Br Med J (Clin Res Ed). 1986 Feb 1;292(6516):344. doi: 10.1136/bmj.292.6516.344. No abstract available. PMID 3080166
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Chandra A, Vaduganathan M, Lewis EF, Claggett BL, Rizkala AR, Wang W, Lefkowitz MP, Shi VC, Anand IS, Ge J, Lam CSP, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Redfield MM, Rouleau JL, Van Veldhuisen DJ, Zannad F, Zile MR, McMurray JJV, Solomon SD; PARAGON-HF Investigators. Health-Related Quality of Life in Heart Failure With Preserved Ejection Fraction: The PARAGON-HF Trial. JACC Heart Fail. 2019 Oct;7(10):862-874. doi: 10.1016/j.jchf.2019.05.015. Epub 2019 Jul 10. PMID 31302043
- [Background] Galinier M, Roubille F, Berdague P, Brierre G, Cantie P, Dary P, Ferradou JM, Fondard O, Labarre JP, Mansourati J, Picard F, Ricci JE, Salvat M, Tartiere L, Ruidavets JB, Bongard V, Delval C, Lancman G, Pasche H, Ramirez-Gil JF, Pathak A; OSICAT Investigators. Telemonitoring versus standard care in heart failure: a randomised multicentre trial. Eur J Heart Fail. 2020 Jun;22(6):985-994. doi: 10.1002/ejhf.1906. Epub 2020 Jun 15. PMID 32438483
- [Background] Nolte K, Herrmann-Lingen C, Wachter R, Gelbrich G, Dungen HD, Duvinage A, Hoischen N, von Oehsen K, Schwarz S, Hasenfuss G, Halle M, Pieske B, Edelmann F. Effects of exercise training on different quality of life dimensions in heart failure with preserved ejection fraction: the Ex-DHF-P trial. Eur J Prev Cardiol. 2015 May;22(5):582-93. doi: 10.1177/2047487314526071. Epub 2014 Mar 13. PMID 24627449
- [Background] Giuliano C, Karahalios A, Neil C, Allen J, Levinger I. The effects of resistance training on muscle strength, quality of life and aerobic capacity in patients with chronic heart failure - A meta-analysis. Int J Cardiol. 2017 Jan 15;227:413-423. doi: 10.1016/j.ijcard.2016.11.023. Epub 2016 Nov 7. PMID 27843045
- [Background] Peyre H, Leplege A, Coste J. Missing data methods for dealing with missing items in quality of life questionnaires. A comparison by simulation of personal mean score, full information maximum likelihood, multiple imputation, and hot deck techniques applied to the SF-36 in the French 2003 decennial health survey. Qual Life Res. 2011 Mar;20(2):287-300. doi: 10.1007/s11136-010-9740-3. Epub 2010 Oct 1. PMID 20882358